CLINICAL TRIAL: NCT04593576
Title: Effects of Outdoor Sports Activities on Pragmatic Language Skills for Children With Autism in Pakistan.
Brief Title: Impact of Sports Activity on Pragmatic Skills of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00807 Saman Javaid
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Autistic Disorder of Childhood Onset With Full Syndrome
Keywords: outdoor sports; physical activity; communication skills
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured physical activity/outdoor sports. (Experimental): Out door sports and structured physical activity protocol will be administered on children with Autism.
  Interventions: Other: Physical activity protocol/out door sports
- Intensive table teaching control group (Active Comparator): Control group will only be exposed to intensive table teaching instead of physical activity protocol.
  Interventions: Other: Intensive table teaching speech therapy

INTERVENTIONS:
Other: Physical activity protocol/out door sports — Warm up exercise will be administered for 10 minutes, then one-to-five small group of instruction based activity will be administered for 15 minutes. After this whole group will be engaged in ball exercise and cooperative ball games for 20 minutes. At the end cool down and reward activity will be done with participants for 15v minutes.
  Total 1 hour physical activity protocol will be administered twice a week.
  Arms: Structured physical activity/outdoor sports.
Other: Intensive table teaching speech therapy — Control group participants will be given speech therapy session based on intensive table teaching for 30 minutes twice a week.
  Arms: Intensive table teaching control group

SUMMARY:
To investigate the effects of structured physical exercises/outdoor sports on social interaction/communication skills of children with Autism in Pakistan.

DETAILED DESCRIPTION:
The word Autism is derived from the Latin word "Autos'' which means "self" - immersion in one's own world. Autism is a disorder that manifests itself in early childhood, is disabling in many cases and is characterized by severe deficits in communication, social interaction, speech/language delays, sensory issues, repetitive and stereotyped behavior, limited interests. Autism was first described as a disease, by an American physician; Autism later came to be known as ASD (Autism spectrum Disorder) due to numerous disorders, various combinations of disorders, multiple unknown etiologies, subtypes and dynamics of the evolving disease. Autism is on the rise with a prevalence rate of 1-2% of infant population. In 2014, the 67th World Health assembly passed a resolution for "Comprehensive and Co-ordinated efforts for the management of the Autism Spectrum Disorders "which was supported by 60 countries, showing the relevance of the pathology. Research on Autism has increased recently, and publications have nearly doubled in the last 5 years, as this spectrum of disorders continues to baffle doctors and scientists and has no cure till now, but can only be managed.

Benefits of physical exercises/sports have been researched, discussed and documented in great detail in the past. But the purpose of this research study is to explore the (Pragmatic communication and social interaction) benefits of specific sports/physical exercises for children aged 5-7 years who are on the spectrum, children with ASD diagnosis. Psychiatrists maintain that certain brain connections develop in ASD children if they regularly indulge / participate in particular sports like athletics (running, jogging, other track events), hiking (exposure to nature), swimming, cycling, horse- back riding, team sports like; basketball, soccer etc. The co-ordination between right and left sides of the body is more important in these sports. Team sports are also a great way of involving ASD children in a social situation where they are more receptive to learning communication skills while opening up with peers, in a relaxed and happy environment. Endorphin; a neurotransmitter, is released in our body during exercise, which triggers a positive/happy feeling, making ASD children more receptive to learning / acquiring new skills through this mode of intervention.

Since all ASD children are unique, it is important to find the right choice of physical exercise/sport that fits their particular profile/symptoms, biomechanics for this mode of intervention to be effective in improving their pragmatic communication skills and social interaction.

The study aims to research the positive effects of outdoor sports activities on pragmatic language skills development amongst the Autistic children aged 5-7 years in Pakistani population. It will help establish a great mode of therapeutic intervention for developing Pragmatic language skills amongst children with Autism. Once established, this mode of intervention will also assist in creating a platform for much needed community based recreational activities for the Autism families in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students with Autism (mild-moderate)
* Participants will be screened on short sensory profile, fulfilling the criteria of typical performance and probable difference will be included.

Exclusion Criteria:

* individuals with Autism along with any comorbid condition.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Social Interaction tasks ABLLS-R (Assessment of basic language learning Skills-Revised) | 15 days
  Changes from baseline, It provides a comprehensive review of the social interaction. It has 34 tasks having 0-4 scoring. Minimum score is 0 and maximum score is 134.
  It provides a comprehensive review of areas including language, social interaction, self-help, academic and motor skills. The task items within each skill area are arranged from simpler to more complex tasks. Social Interaction comprises of 34 tasks that would be used as a measuring tool in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Zubair, MS-SLP/T, Principal Investigator — Riphah International University
Locations (1):
- Profiles, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fedotchev AI, Dvoryaninova VV, Velikova SD, Zemlyanaya АА. Modern Technologies in Studying the Mechanisms, Diagnostics, and Treatment of Autism Spectrum Disorders. Современные технологии в медицине. 2019;11(1 (eng)).
- [Background] Tse CYA, Pang CL, Lee PH. Choosing an Appropriate Physical Exercise to Reduce Stereotypic Behavior in Children with Autism Spectrum Disorders: A Non-randomized Crossover Study. J Autism Dev Disord. 2018 May;48(5):1666-1672. doi: 10.1007/s10803-017-3419-3. PMID 29196864
- [Background] Zhao M, Chen S. The Effects of Structured Physical Activity Program on Social Interaction and Communication for Children with Autism. Biomed Res Int. 2018 Jan 15;2018:1825046. doi: 10.1155/2018/1825046. eCollection 2018. PMID 29568743
- [Background] DAN YJ, SU LY, LIU YH. Case Study on PE Intervention of the Communicative Behaviors of Autistic Infants [J]. Journal of Tianjin University of Sport. 2006;2. (Article in Chinese)
- [Background] MA K. Examining the perceived impacts of recreational swimming lessons for children with autism spectrum disorder. International Journal of Aquatic Research and Education. 2019;10(4):6.
- [Background] Cei A, Franceschi P, Rosci M, Sepio D, Ruscello B. Motor and psychosocial development in children with autism spectrum disorder through soccer. International Journal of Sport Psychology. 2017;48(5):485-507.
- [Background] Howells K, Sivaratnam C, Lindor E, Hyde C, McGillivray J, Whitehouse A, Rinehart N. Can Participation in a Community Organized Football Program Improve Social, Behavioural Functioning and Communication in Children with Autism Spectrum Disorder? A Pilot Study. J Autism Dev Disord. 2020 Oct;50(10):3714-3727. doi: 10.1007/s10803-020-04423-5. PMID 32107700
- [Background] Howells K, Sivaratnam C, May T, Lindor E, McGillivray J, Rinehart N. Efficacy of Group-Based Organised Physical Activity Participation for Social Outcomes in Children with Autism Spectrum Disorder: A Systematic Review and Meta-analysis. J Autism Dev Disord. 2019 Aug;49(8):3290-3308. doi: 10.1007/s10803-019-04050-9. PMID 31102193
- [Background] Yu CCW, Wong SWL, Lo FSF, So RCH, Chan DFY. Study protocol: a randomized controlled trial study on the effect of a game-based exercise training program on promoting physical fitness and mental health in children with autism spectrum disorder. BMC Psychiatry. 2018 Feb 27;18(1):56. doi: 10.1186/s12888-018-1635-9. PMID 29486750